CLINICAL TRIAL: NCT02073955
Title: Adaptation and Validation of a Community Worker Administered Stroke Symptom Questionnaire in a Peri-urban Pakistani Community
Brief Title: Validation of a Community Worker Administered Stroke Symptom Questionnaire
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor, Aga Khan University
Other Study IDs: 5D43TW008660-02 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
Keywords: Stroke; Validation; Community Health workers; stroke symptom questionnaire
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pakistani adults: Men and women aged 40 and above, residing in Ibrahim Hyderi (periurban Pakistani community)
  Consenting to Interview about stroke symptoms

SUMMARY:
This is a validation study. A stroke symptom questionnaire will be adapted and translated into local language. Two community health workers will be trained in its administration. Their findings will be validated against assessment by two neurologists.

The study hypothesis is that the chance corrected agreement between the community worker administered stroke symptom questionnaire and the assessment by neurologist based on history and physical examination is at least moderate.

DETAILED DESCRIPTION:
Overall Objective: To translate, adapt and validate a stroke symptom questionnaire for identification of stroke symptoms by community health workers ( CHW) in a peri-urban Pakistani community

Specific Aims:

1. To translate and adapt a stroke symptom questionnaire for identification of stroke symptoms by community workers in a peri-urban Pakistani community
2. To validate community workers administered stroke symptom questionnaire against assessment by neurologist in a peri-urban Pakistani community
3. To determine the feasibility of utilizing community workers for identification of stroke patients in the community in terms of subject refusals and difficulty in understanding questions

The study will be conducted at the community site of AMAN community health project in Ibrahim Hyderi. Community health workers will systematically select households and from them individuals meeting eligibility criteria will be interviewed. Community workers will administer stroke symptom questionnaire to them at their homes. Those unable to answer will have a surrogate answering for them. In the second part of the study, two neurologists will independently assess all individuals. The purpose of this would be to validate the findings of the community workers based on the stroke symptom questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 and above
* Permanent resident of Ibrahim Hyderi
* All ethnicities
* Can answer for themselves or have a surrogate willing to provide necessary information. Surrogate is defined as one who lives in the same household as the individual, who is the primary caregiver and has access to the medical record / information of the patient.
* Willing to give written informed consent

Exclusion Criteria:

- Individuals refusing to participate in any of the two components of the study i.e. CHW interview or neurological assessment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (above 40 years of age) residing in Ibrahim Hyderi and willing to participate in the all components of the study
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Validity | Cross-sectional , All interviews within 4 Weeks ( CHW and Neurologist)
  This was a validation study in which we calculated the sensitivity, specificity and predictive values for CHW administered questionnaire against assessment by two neurologists. We also assessed the chance corrected agreement (kappa) for the same.

SECONDARY OUTCOMES:
Feasibility | Cross sectional - All interviews within 4 weeks( CHW and Neurologists)
  We assessed the feasibility of utilizing CHWs for stroke screening in terms of time taken to fill out questionnaire, difficulty in understanding questions and subject refusals

OTHER OUTCOMES:
Prevalence of stroke symptoms | Cross-sectional _ All interviews within 4 weeks, by CHWS using validated questionairre
  Once validated, we used the CHW administered tool to assess stroke symptom prevalence in this community

CONTACTS AND LOCATIONS:
Overall Officials: Ayeesha K Kamal, Study Director — AKUH; Maria Khan, Principal Investigator — AKUH
Locations (1):
- Community Health Center, Ibrahim Hyderi, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Khan M, Kamal AK, Pasha O, Islam M, Azam I, Virk A, Nasir A, Andani A, Jan M, Akhtar A, Razzak JA. Study Protocol: Validation and Adaptation of community-worker-administered stroke symptom questionnaire in a periurban Pakistani community to determine disease burden. J Vasc Interv Neurol. 2015 Feb;8(1):1-10. PMID 25825625